CLINICAL TRIAL: NCT03001739
Title: Intensive Blood PRessure Control in Patients With Acute Type B AortIc Dissection (RAID): Study Protocol for Randomized Controlled Trial
Brief Title: Intensive Blood PRessure Control in Patients With Acute Type B AortIc Dissection
Acronym: RAID
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Jian-cang Zhou M.D., Principal Investigator, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160920-9
Record Dates: First submitted 2016-12-10; First posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Blood High Pressure; Aortic Dissection Type B
MeSH Terms: conditions — Hypertension | interventions — urapidil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive BP control (<120mmHg) (Experimental): Urapidil Hydrochloride Injection (100-400ug/min) or other antihypertensive agents to decrease the BP to < 120 mm Hg
  Interventions: Drug: Urapidil Hydrochloride Injection
- Conventional BP control (120-140mmHg) (Active Comparator): Urapidil Hydrochloride Injection (100-400ug/min) or other antihypertensive agents to decrease the BP to 120-140 mm Hg
  Interventions: Drug: Urapidil Hydrochloride Injection

INTERVENTIONS:
Drug: Urapidil Hydrochloride Injection — Urapidil Hydrochloride Injection or other antihypertensive agents to decrease the BP to the target level.
  Other Names: Urapidil

SUMMARY:
Aortic dissection (AD) aneurysm is a common catastrophic aortic disease in clinical setting. Conservative therapy of heart rate and blood pressure control in the acute phase is the essential treatment as guidelines recommended. Nevertheless, there is no unanimous optimal target for blood pressure in patients with AD so far. The American Heart Association and the Canadian Cardiovascular Society recommend the blood pressure should be controlled to lower than 140/90mmHg, while for patients with diabetes or chronic renal failure, the blood pressure target should be no less than 130/80 mmHg. Recently, the Japanese Circulation Society recommended that the blood pressure should be controlled to no less than 130mmHg. However, there was few large-scale, randomized, controlled studies reported on the effect of different blood pressure control levels on the prognosis of patients with AD. Hence, the intensive control of blood pressure to <120 mmHg, compared to <140 mmHg, may improve the patients' outcome. Thus, in this study, the effect of intensive blood pressure control (<120mmHg) with conventional blood pressure control (<140mmHg) on the prognosis of ABAD patients will be compared, and to identify the therapeutic efficacy of intensive blood pressure control on the ABAD patients.

DETAILED DESCRIPTION:
Aortic dissection (AD) aneurysm is a common catastrophic aortic disease in clinical setting. In the U.S., the prevalence is approximate 2.9-3.5 cases/100000 persons per year, with recent evidence showing an increasing incidence of up to 14 cases per 100000 patients per year. AD aneurysm can be classified into the types of Stanford A and B based on whether the ascending aorta was being involved. For acute type B aortic dissection (ABAD), which is generally accounted for one thirds of all aortic dissection and is especially more common among Chinese due to the suboptimal control of blood pressure. Optimal treatment of ABAD from symptom onset remains uncertain. Conservative therapy of heart rate and blood pressure control in the acute phase is the essential treatment for patient without serious complications such as concurrent mesenteric artery or lower limb arterial embolism. The long-term survival of ABAD is still low though great improved in medication optimization and surgical repair technique in the past decades. It was reported that 5-year and 10-year survival rates for ABAD were 60% and 35% respectively. As the development of minimally invasive techniques in recent years, the endovascular repair procedure has become a routine procedure in the treatment of patient with ABAD, this rendered an improved prognosis with a 5-year survival rate close to 80%.

Hypertension is well known as the most common cause for AD. The statistics from International Registry of Acute Aortic Dissection (IRAD) demonstrated that 72.1% of AD patients had a history of hypertension. The hypertension may aggravate hematoma expansion and results in serious consequences. Therefore, effectively blood pressure control may alleviate the severe pain caused by acute AD and lessen the progression of arterial dissection. The control of hypertension is the primary treatment for acute aortic dissection, and should be maintained throughout the entire treatment. Currently, all guidelines recommended to decline the transaortic pressure via controlling the heart rate and blood pressure for AD patient in acute phase. Theoretically, to control the blood pressure to the minimal level meeting the sufficient end-organ perfusion can decrease the risk of vessel rupture as much as possible. Whereas, too much low blood pressure target may increase the mortality of patients. Powell and his colleague found when the minimum blood pressure increased by 10mmHg (vs. <70 mmHg, maximal to 120 mmHg) for AD patients, the risk of death decreased by 12% (OR = 0.88, P <0.001).

Nevertheless, there is no unanimous optimal target for blood pressure in patients with AD so far. The American Heart Association and the Canadian Cardiovascular Society recommend the blood pressure should be controlled to lower than 140/90mmHg, while for patients with diabetes or chronic renal failure, the blood pressure target should be no less than 130/80 mmHg. Recently, the Japanese Circulation Society recommended that the blood pressure should be controlled to no less than 130mmHg. Hence, the intensive control of blood pressure to <120 mmHg, compared to <140 mmHg, may improve the patients' outcome. Thus, in this study, the effect of intensive blood pressure control (<120mmHg) with conventional blood pressure control (<140mmHg) on the prognosis of ABAD patients will be compared.

Methods Study design and setting The study was a prospective randomized controlled trial that will recruit a maximal of 360 patients in eight tertiary Chinese hospitals over 2 years. All patients with new diagnosed ABAD in the participating hospitals will be screened for potential eligibility. The study was approved by the ethics committee of the hospitals (20160920-9). Written informed consents will be signed by the patients or their legally authorized representatives. The study was registered in the website of ClinicalTrial.gov .

Sites and patients Doctors from eight hospitals attended the kick-off meeting held in Courtyard Marriott, Hangzhou, March 19th, 2016, and discussed the research protocol and details. The amended research protocol was passed according to revised discussion results and the agreement of all participating units. The methods of blood pressure measurement and the apparatus used are unified. All hospitals will adopt similar non-invasive blood pressure monitoring method and unified monitoring frequency to observe whether the blood pressure is controlled within the target range in two groups. Likewise, the blood pressure target after discharge was maintained at the same levels.

All patients with AD from the participating hospitals who conform to the following inclusion and exclusion criteria will be randomized. Inclusion and exclusion criteria were shown in other parts.

Randomization Blocked randomization was adopted and the intensive and conventional blood pressure control treatments were allocated at random in a ratio of 1:1 in blocks of sizes of 4,6,8, and 10 to 360 subjects. The study is an open label trial. After investigators in each participating centers screened the potential patients within 4 hours after acute onset, a number from a pre-allocated envelope will be gotten and which denotes which group the patient will be allocated to.

Treatments All the patients were admitted to ICU or general wards at the discretion of doctors. Based on the guidelines of aortic management, all patients received analgesic therapy and standard control of heart rate and blood pressure treatments. Intravenous esmolol was used for continuous control of heart rates. Choice of intravenous antihypertensive agents was at the discretion of the in charge physicians. After the stabilization of the situation, the intravenous medications were shifted to the oral treatments. The target blood pressure for the intensive and conventional groups were <140mmHg and <120mmHg respectively. For most patients, they will undergo an endovascular treatment approximate two weeks later.

Study endpoints The primary outcome is a composite in-hospital adverse outcome, including death, permanent paraplegia or semi- paralysis during the hospitalization, and renal failure requiring hemodialysis at discharge.

The secondary outcomes include the mortality in 6-month and 1-year, ICU length of stay, total length of hospital stay, postoperative renal injury, and re- intervention.

Data collection Research coordinators of individual participating hospital will collect the required data on the case report form. However, the data was de-named and special security code was required to access the data. To facilitate the communications between investigators, the case report form was written in Chinese. The primary research institute is responsible for collecting and checking the data of all centers; and will contact the co-investigators in various centers for checking or revising should they had any question. The primary research institute has established an independent study quality control group to implement the disposal plan for all unexpected circumstances that may occur.

Sample size calculation and interim analysis The primary outcome was a composite in-hospital adverse outcome, including the death, stroke, permanent paraplegia or semi- paralysis during the hospitalization, and renal failure requiring hemodialysis at discharge. Bashir et al reported that the incidence of comprehensive nosocomial severe prognostic adverse events of ABAD was 45.2%. Assume that the incidence of severe prognosis adverse event in comprehensive hospital after intensive blood pressure control could be reduced to 30%, so a total of 322 subjects enrolled in the study are sufficient to find the difference statistically between two groups through the appropriate software calculation under the power of 0.8 and at the two-side test with α = 0.05. Considering a dropout rate of 10%, it is proposed to include 360 cases totally into the study. A formal interim analysis was conducted halfway during study enrollment. The overall type I error was controlled using an O'Brien-Fleming spending function, with a final significance level of 0.05 for the primary end point.

Statistical analysis Descriptive data were reported as either mean ± SD, median (interquartile range) or number and percentage. With respect to the differences between two groups, categorical variables were compared using chi-square analysis. Continuous variables were compared using Independent Sample T test for normally distributed data and Mann-Whitney U test for non-normally distributed data. For survival analyses, Kaplan-Meier estimates were generated to assess differences between groups using the log-rank test, and expressed the data as cumulative mortality curves. Statistical analysis was performed by using SPSS 16.0 (Chicago, Ill, USA) and PASS 11.0. Statistical significance was defined as a P value <0.05.

Discussion ABAD comprises approximately 30% of all aortic dissection cases. In contrast with type A aortic dissection, patients with type B dissection are tend to be older, have higher rates of atherosclerosis. Initial goals for acute aortic dissection management are directed at control of blood pressure and heart rate, which subsequently limiting propagation of the false lumen by controlling aortic shear stress. Whilst medical management has demonstrated an in-hospital mortality rate less than 10%, post-discharge the acute type B aortic disease continues to evolve eventually resulting in complicated type B disease. Moreover, complicated acute type B aortic dissection shows even more striking mortality as high as 30%, particularly in the elderly. Poor control of blood pressure was believed to be one of the main reasons for the progress of the type B aortic dissection into complications or even the laceration extended to the ascending aorta. Dalsart and colleague demonstrated that a systolic blood pressure more than 130 mmHg was associated with a bigger aortic enlargement in type B aortic dissection (P=0.02) . In another study of 25 years follow-up in 252 patients who received repair of acute type A aortic dissection, patients who maintained a systolic blood pressure <120 mm Hg had improved freedom from reoperation, compared to those target blood pressure 120-140 mm Hg or >140 mm Hg. Hence, most guidelines recommended a reasonable initial target for systolic blood pressure is between 100 and 120 mm Hg. However, this target is based on the hypothesis that all the end-organs blood supply is not compromised. Data from International Registry of Acute Aortic Dissection (IRAD) has shown that approximately one quarter of patients presenting with acute type B aortic dissection are followed into complicated category, including malperfusion of spinal arteries leading to paresis, and paraplegia or malperfusion of visceral arteries leading to abdominal pain. Thus, how to balance the decrease of blood pressure to the lowest amount and maintain adequate end-organ perfusion is a challenge. Given vast majority patients with type B aortic dissection had a history of hypertension, a too lower target of blood pressure may comprise the cerebral perfusion or complicated organ perfusion, which consequently caused stroke or other morbidity such as ischemic intestinal necrosis. On the other hand, a much strict blood pressure target and sometimes constrain on the patients daily activities may aggravate patients' worry, which inversely increased increase the blood pressure. Unfortunately, there is no empirical data or trials to guide the optimal blood pressure target setting for various patients. Hence, the study was designed to bridge the gap.

In conclusion, the investigators believe that the study will provide new insight into the of blood pressure management of patients of acute Type B aortic dissection and subsequently improve the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with Stanford type B acute aortic dissection and systolic blood pressure>160mmHg

Exclusion Criteria:

* Age <18 years,
* In pregnancy,
* Diagnosis of aortic dissection was made 48 hours or more prior,
* Dissection due to aortic intramural hematoma or penetrating atherosclerotic ulcer,
* With history of previous surgical or interventional endovascular treatment for aortic diseases,
* With traumatic aortic injury,
* With history of cerebrovascular accident, brain surgery, chronic renal insufficiency, and mesenteric vascular thrombosis or dissection,
* AD patient concomitant with new cerebral infarction, or ischemic mesenteric artery or lower limb arteries which requiring urgent surgical interventions,
* With obvious contraindications for antihypertensive therapy, such as severe carotid stenosis, cerebral infarction in acute phase ,
* Pathogenesis of the dissection was due to congenital aortic hypoplasia, such as Marfan syndrome, connective tissue diseases.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
composite in-hospital adverse outcome | From date of randomization until the date of death from any cause，or permanent paraplegia or semi- paralysis during the hospitalization, and renal failure requiring hemodialysis at discharge, whichever came first, assessed up to 3 months
  including death, permanent paraplegia or semi- paralysis during the hospitalization, and renal failure requiring hemodialysis at discharge

SECONDARY OUTCOMES:
mortality | 6-month and 1-year after onset of the dissection
  All cause mortality
ICU length of stay | From date of ICU admission until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 3 months
re-operation or another endovascular intervention for the same problem | From date of first intervention until the date of second intervention, assessed up to 12 months
  any intervention for the same situation such as operation or endovascular intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yun-song Yu, MD, Study Director — Zhejiang University
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou JC, Zhang N, Zhang ZH, Wang TT, Zhu YF, Kang H, Zhang WM, Li DL, Li WD, Liu ZJ, Qian XM, Zhang MY, Wang J, Zhou M, Yang ZT, Yu YX, Li HY, Zhang J, Wang YG, Gao JP, Ling L, Pan KH; Pressure in Acute Type B Aortic Dissection (RAID) study group. Intensive blood pressure control in patients with acute type B aortic dissection (RAID): study protocol for randomized controlled trial. J Thorac Dis. 2017 May;9(5):1369-1374. doi: 10.21037/jtd.2017.03.180. PMID 28616291